CLINICAL TRIAL: NCT01698762
Title: IADAPT-Third Phase
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2012-0172; 1R18HS019354-02 (AHRQ); NCI-2016-00638 (Registry Identifier: NCI-CTRP)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Musculoskeletal Diseases
Keywords: Musculoskeletal Diseases; Osteoarthritis; OA; Rheumatoid Arthritis; RA; Osteoporosis; OP; Multimedia Patient Decision Aids; MM-PtDAs; DVD; Comparative Effectiveness Research Summary Guide; CERSG; Booklet; Questionnaires; Surveys
MeSH Terms: conditions — Musculoskeletal Diseases; Osteoarthritis; Arthritis, Rheumatoid; Osteoporosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Osteoarthritis (OA): One OA group will watch a DVD - Multimedia Patient Decision Aids (MM-PtDAs) of information about their disease type.
  One OA group will read a booklet - Comparative Effectiveness Research Summary Guide (CERSG) about their disease type.
  Questionnaires completed at baseline, 3, and at 6 months.
  Interventions: Other: Multimedia Patient Decision Aids (MM-PtDAs); Other: Comparative Effectiveness Research Summary Guide (CERSG); Behavioral: Questionnaires
- Osteoporosis (OP): One OP group will watch a DVD - Multimedia Patient Decision Aids (MM-PtDAs) of information about their disease type.
  One OP group will read a booklet - Comparative Effectiveness Research Summary Guide (CERSG) about their disease type.
  Questionnaires completed at baseline, 3, and at 6 months.
  Interventions: Other: Multimedia Patient Decision Aids (MM-PtDAs); Other: Comparative Effectiveness Research Summary Guide (CERSG); Behavioral: Questionnaires
- Rheumatoid Arthritis (RA): One RA group will watch a DVD - Multimedia Patient Decision Aids (MM-PtDAs) of information about their disease type.
  One RA group will read a booklet - Comparative Effectiveness Research Summary Guide (CERSG) about their disease type.
  Questionnaires completed at baseline, 3, and at 6 months.
  Interventions: Other: Multimedia Patient Decision Aids (MM-PtDAs); Other: Comparative Effectiveness Research Summary Guide (CERSG); Behavioral: Questionnaires

INTERVENTIONS:
Other: Multimedia Patient Decision Aids (MM-PtDAs) — Patient group will watch a DVD of information about their disease type.
  Other Names: DVD
Other: Comparative Effectiveness Research Summary Guide (CERSG) — Patient group to read a booklet about their disease type.
  Other Names: Booklet; Reading material
Behavioral: Questionnaires — Questionnaires completed at baseline, 3, and at 6 months.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to compare a booklet and a DVD for patients with knee osteoarthritis, osteoporosis, or rheumatoid arthritis.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups:

* Group 1 will watch a DVD and receive a booklet of information about their disease type (knee osteoarthritis, osteoporosis, or rheumatoid arthritis).
* Group 2 will read a booklet about their disease type.

All the materials including the DVD, booklet, and questionnaires will be in English and Spanish. You may choose which language you prefer to use while watching and/or reading the materials.

You will be asked to complete questionnaires before and after watching the DVD or reading the booklet. We will ask you about how the material made you think and feel and how easy or hard the material was to understand.

You will also fill out short questionnaires that include questions about your demographic information, your health, your thoughts about bone/joint disease, how you might choose treatments for bone/joint disease, and how you make treatment decisions. These questionnaires will take up to 45 minutes to complete in the clinic.

This first visit will take about 60-90 minutes total to complete. If you are unable to complete this first visit today you will need to complete it within the next two weeks.

You will be asked to fill out these questionnaires again 3 months and 6 months later, by mail. The study staff will mail you the questionnaires, along with a postage-paid return envelope that you can use to send the questionnaires back. If you prefer you can also complete the questionnaires over the phone or the research staff can meet you at the clinic or your home to complete the questionnaires at 3 and 6 months.

Your participation on this study will be over after you have mailed back the 6-month questionnaires.

This is an investigational study.

Up to 828 participants will take part in this multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. Knee Osteoarthritis (OA): (a) age 45 and over (b) prior diagnosis of knee OA (unilateral or bilateral) by a physician.
2. Rheumatoid Arthritis (RA): (a) age 18 and over, (b) compliance with American College of Rheumatology criteria for the diagnosis of RA, (c) and disease duration < or = 10 years
3. Osteoporosis (OP): (a) female gender, (b) age 45 and over, (c) and at least 3 years post-menopausal
4. Adequate cognitive status as determined by the research assistant (see description in "Recruitment Eligibility")
5. Ability to communicate in English or Spanish language without a translator
6. Have access to a telephone

Exclusion Criteria:

1. Hospitalized
2. Patients with RA or knee OA who also have any other connective tissue disease or spondyloarthropathy.
3. Patients with diagnosis of RA and disease duration (>10 years)
4. Patients who do not sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Harris County Hospital District (HCHD) and Kelsey-Seybold patients in rheumatology, internal medicine and family practice clinics.
Sampling Method: Non-Probability Sample
Enrollment: 676 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Disease Knowledge and Therapeutic Options | 3 months
  Primary analyses performed using repeated measures ANOVA, with group allocation - multimedia patient decision aids (MM-PtDA) vs. Comparative Effectiveness Research Summary Guide (CERSG) as the factor of interest and knowledge as the central outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Angeles M. Lopez-Olivo, MD, PHD, MS, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Kelsey-Seybold Clinic, Houston, Texas
  - Harris County Hospital District (HCHD), Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Lopez-Olivo MA, des Bordes JKA, Jibaja-Weiss M, Volk RJ, Suarez-Almazor ME. Preferred Strategies for Delivering Health Information to Patients With Musculoskeletal Disorders: A Qualitative Study. J Clin Rheumatol. 2022 Jan 1;28(1):e102-e109. doi: 10.1097/RHU.0000000000001627. PMID 33298811
- [Background] Lopez-Olivo MA, Ingleshwar A, Volk RJ, Jibaja-Weiss M, Barbo A, Saag K, Leong A, Suarez-Almazor ME. Development and Pilot Testing of Multimedia Patient Education Tools for Patients With Knee Osteoarthritis, Osteoporosis, and Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2018 Feb;70(2):213-220. doi: 10.1002/acr.23271. Epub 2017 Dec 29. PMID 28464546
- [Background] Lopez-Olivo MA, Lin H, Rizvi T, Barbo Barthel A, Ingleshwar A, des Bordes JKA, Jibaja-Weiss M, Volk RJ, Suarez-Almazor ME. Randomized Controlled Trial of Patient Education Tools for Patients With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2021 Oct;73(10):1470-1478. doi: 10.1002/acr.24362. Epub 2021 Aug 31. PMID 32583971
- [Background] Lopez-Olivo MA, des Bordes JK, Lin H, Volk RJ, Rizvi T, Suarez-Almazor ME. A Randomized Controlled Trial Comparing Two Self-Administered Educational Strategies for Patients With Knee Osteoarthritis. ACR Open Rheumatol. 2021 Mar;3(3):185-195. doi: 10.1002/acr2.11222. Epub 2021 Feb 16. PMID 33590950
- [Background] Lopez-Olivo MA, des Bordes JKA, Lin H, Rizvi T, Volk RJ, Suarez-Almazor ME. Comparison of multimedia and printed patient education tools for patients with osteoporosis: a 6-month randomized controlled trial. Osteoporos Int. 2020 May;31(5):857-866. doi: 10.1007/s00198-019-05210-4. Epub 2019 Dec 16. PMID 31844906
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org